CLINICAL TRIAL: NCT05615363
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Doseranging Trial of OPC-131461 in Cardiac Edema (Congestive Heart Failure [CHF])
Brief Title: A Dose-ranging Trial of OPC-131461 in Cardiac Edema (Congestive Heart Failure [CHF])
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 351-102-00004; jRCT (Registry Identifier: jRCT2071220069)
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Edema (CHF)
MeSH Terms: conditions — Edema, Cardiac; Heart Failure | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- OPC 131461 10mg group (Experimental): OPC-131461 5 mg tablet ｘ 2
  Interventions: Drug: OPC 131461 10mg group
- OPC 131461 5mg group (Experimental): OPC-131461 5 mg tablet and placebo tablet
  Interventions: Drug: OPC 131461 5mg group
- OPC 131461 2mg group (Experimental): OPC-131461 1 mg tablet ｘ 2
  Interventions: Drug: OPC 131461 2mg group
- OPC 131461 1mg group (Experimental): OPC-131461 1 mg tablet and placebo tablet
  Interventions: Drug: OPC 131461 1mg group
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPC 131461 10mg group — OPC-131461 5 mg tablet x 2，once-daily oral administration for 14 days
  Arms: OPC 131461 10mg group
Drug: OPC 131461 5mg group — OPC-131461 5 mg tablet and placebo tablet，once-daily oral administration for 14 days
  Arms: OPC 131461 5mg group
Drug: OPC 131461 2mg group — OPC-131461 1 mg tablet x 2，once-daily oral administration for 14 days
  Arms: OPC 131461 2mg group
Drug: OPC 131461 1mg group — OPC-131461 1 mg tablet and placebo tablet，once-daily oral administration for 14 days
  Arms: OPC 131461 1mg group
Drug: Placebo — Placebo tablet，once-daily oral administration for 14 days
  Arms: Placebo

SUMMARY:
To investigate the dose response in respect of weight decrease following repeated oral administration of OPC-131461 at 1, 2, 5, and 10 mg or placebo in patients with CHF with volume overload despite having received diuretics other than vasopressin antagonists

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CHF with lower limb edema, pulmonary congestion, or jugular venous distension due to volume overload.
* Subjects undergoing any of the following diuretic therapies

  * Loop diuretics at a dosage equivalent to 40 mg/day or more of furosemide tablet/fine granule
  * Concomitant administration of a loop diuretic and a thiazide diuretic (including similar drugs) at any doses
  * Concomitant administration of a loop diuretic and a mineralocorticoid receptor antagonist or potassium-sparing diuretic at any doses
* Subjects who were currently hospitalized or who are able to be hospitalized

Exclusion Criteria:

* Subjects with acute heart failure
* Subjects with an assisted circulation device
* Subjects who cannot sense thirst or who have difficulty in ingesting water

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Tsunoda, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Harasanshin Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Groups:
- Material A: OPC 131461 10mg group
- Material B: OPC 131461 5mg group
- Material C: OPC 131461 2mg group
- Material D: OPC 131461 1mg group
- Placebo: Placebo
Period: Overall Study
Arm/Group | Material A | Material B | Material C | Material D | Placebo
Started | 31 | 32 | 31 | 33 | 30
Completed | 27 | 28 | 22 | 29 | 25
Not Completed | 4 | 4 | 9 | 4 | 5
Not completed — Adverse Event | 0 | 4 | 4 | 3 | 1
Not completed — Physician Decision | 2 | 0 | 4 | 1 | 3
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set, which included all randomized patients who received ≥1 dose of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Material A | Material B | Material C | Material D | Placebo | Total
Number analyzed (Participants) | 31 | 32 | 31 | 33 | 30 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 3 | 3 | 5 | 22
  >=65 years | 25 | 27 | 28 | 30 | 25 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.5 (11.6) | 75.2 (10.7) | 75.3 (13.1) | 76.7 (7.9) | 76.4 (9.4) | 75.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 2 | 11 | 12 | 58
  Male | 17 | 13 | 29 | 22 | 18 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 31 | 32 | 31 | 33 | 30 | 157
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight From Baseline to Last Assessment Time Point (the Day After IMP Administration) by Day 8
Description: Calculate the change in body weight from the baseline up to Day 8 (kg)
Time Frame: Baseline, Day 8
Population: The full analysis set includes all subjects who have been administered at least one treatment of the IMP, and for whom efficacy data after IMP administration are available.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Material A | Material B | Material C | Material D | Placebo
Number analyzed (Participants) | 31 | 32 | 31 | 33 | 30
kg | -1.96 [-2.50 to -1.42] | -1.74 [-2.28 to -1.20] | -1.4 [-1.94 to -0.85] | -1.84 [-2.36 to -1.31] | -1.17 [-1.72 to -0.62]

2. Secondary Outcome: Change in Body Weight From Baseline to Last Assessment Time Point (the Day After IMP Administration) by Day 15
Description: Calculate the percentage change in body weight from the baseline up to last assessment time point (the day after IMP administration) by Day 15 （％）
Time Frame: Baseline, Day15
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Material A | Material B | Material C | Material D | Placebo
Number analyzed (Participants) | 31 | 32 | 31 | 33 | 30
kg | -2.12 [-2.80 to -1.44] | -2.11 [-2.79 to -1.43] | -1.72 [-2.41 to -1.03] | -1.87 [-2.53 to -1.21] | -1.38 [-2.07 to -0.69]

3. Secondary Outcome: Improvement of or Change in Congestive Findings ( Lower Limb Edema ) From Baseline to Last Assessment Time Point (the Day of IMP Administration) by Day 7
Description: The tibial margins or acrotarsia in a sitting position will be examined to assess the severity of edema according to the criteria in 0 : Absent, No pitting observed at all, 1:Mild,Slight pitting observed, 2:Moderate, Pitting observed, 3 : Severe,Apparent edema.
  Improvement rates (percentages of subjects who have symptoms at baseline and show markedly improved or improved after IMP administration) and resolution rates (percentages of subjects who have symptoms at baseline and no symptoms after IMP administration) at the last assessment time point (the day of IMP administration) by Day 7.
Time Frame: Baseline, Day7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Material A | Material B | Material C | Material D | Placebo
Number analyzed (Participants) | 22 | 23 | 24 | 24 | 24
Participants | 16 | 18 | 9 | 19 | 19

4. Secondary Outcome: Improvement of or Change in Congestive Findings ( Pulmonary Congestion ) From Baseline to Last Assessment Time Point (the Day of IMP Administration) by Day 7
Description: The severity of pulmonary congestion will be determined according to the criteria in 0 : Absent, No congestion, 1:Mild,Pulmonary venous congestion, 2:Moderate, Interstitial pulmonary edema, 3 : Severe, Alveolar pulmonary edema.
  Improvement rates (percentages of subjects who have symptoms at baseline and show markedly improved or improved after IMP administration) and resolution rates (percentages of subjects who have symptoms at baseline and no symptoms after IMP administration) at the last assessment time point (the day of IMP administration) by Day 7.
Time Frame: Baseline, Day7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Material A | Material B | Material C | Material D | Placebo
Number analyzed (Participants) | 23 | 26 | 20 | 26 | 24
Participants | 21 | 19 | 10 | 22 | 18

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until follow-up for up to 10 - 14 days after the last dose of study medication.
Description: All AEs will be coded by system organ class and MedDRA preferred term. The incidence of the following events will be summarized by treatment group. If the same event occurs more than once in the same subject, the higher severity will be used. TEAEs related to the IMP will be tabulated similarly.
Arm/Group | Material A | Material B | Material C | Material D | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32 | 0/31 | 1/33 | 1/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 2/32 | 0/31 | 1/33 | 1/30
Other Adverse Events (participants affected / at risk) | 11/31 | 8/32 | 12/31 | 14/33 | 8/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Material A (N=31) | Material B (N=32) | Material C (N=31) | Material D (N=33) | Placebo (N=30)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Material A (N=31) | Material B (N=32) | Material C (N=31) | Material D (N=33) | Placebo (N=30)
Constipation (Gastrointestinal disorders) | 2 | 2 | 4 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0
Thirst (General disorders) | 4 | 4 | 0 | 4 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Blood pressure decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 5 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 1 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT05615363/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT05615363/SAP_001.pdf